CLINICAL TRIAL: NCT00387842
Title: A Randomized Clinical Trial Comparing Laparoscopic and Open Surgery for Colon Cancer
Brief Title: COlon Cancer Laparoscopic or Open Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLOR I
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopic surgery
Procedure: Conventional surgery

SUMMARY:
COLOR trial is a randomized, international, multi center study comparing the outcomes of laparoscopic and conventional resection of colon carcinoma with curative intent. Clinical and operative data will be collected centrally in the coordinating centre in Rotterdam, The Netherlands. Quality of life and costs will be assessed on a national basis.

DETAILED DESCRIPTION:
The design involves allocation of all suitable consecutive patients with colon carcinoma to either of the two procedures at a randomization ratio of 1:1. The trial will be stratified according to participating centre, resection type and gender.

Disease free survival for all TNM stages after 3 years is currently about 70%. To detect a difference of 7% in disease free survival rate after 3 years between open and laparoscopic resection of colon cancer, 1200 patients will have to be included (60 vs 67%, two-sided analysis; alfa=0.05, beta=0.20, power=80% and p=0.05). All analyses will be performed on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Solitary colon carcinoma observed at colonoscopy or on barium enema X-ray within 28-days before operation (no biopsy required)
* Polyp containing invasive carcinoma according to colonoscopic biopsy, undertaken within 28 days before operation
* Suitable for elective surgical resection by right hemicolectomy, left hemicolectomy or sigmoid resection
* Sigmoid colon tumour cranially to conjugata diagonalis on lateral view of barium enema
* BMI < 30 kg/m2
* Informed consent according to local requirements

Exclusion Criteria:

* Carcinoma of the splenic flexure
* Carcinoma of the transverse colon
* Signs of acute intestinal obstruction
* More than one colon tumour
* Scheduled need for other synchronous colon surgery
* Synchronous surgery ofr other intra-abdominal organs
* Pre-operative indication of invasion of adjacent organs
* Pre-operative evidence of distant metastases
* Previous ipsilateral colon surgery
* Other malignancies in medical history, except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri
* Absolute contra-indications to general anaesthesia or prolonged pneumoperitoneum, such as severe cardiovascular or respiratory disease
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 1997-03; Study Completion 2008-03

PRIMARY OUTCOMES:
Primary endpoint is cancer free survival at three years.

SECONDARY OUTCOMES:
Secondary endpoints are overall survival at three and five years, 28 day mortality and morbidity, quality of life, costs, location and rates of recurrences and pathologic anatomic characteristics of the resected specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Bonjer, MD, PhD, Principal Investigator — Dalhousie University, CDHA / Erasmus MC Rotterdam

REFERENCES:
- [Derived] Koedam TWA, Bootsma BT, Deijen CL, van de Brug T, Kazemier G, Cuesta MA, Furst A, Lacy AM, Haglind E, Tuynman JB, Daams F, Bonjer HJ; on behalf of the COLOR COLOR II study group. Oncological Outcomes After Anastomotic Leakage After Surgery for Colon or Rectal Cancer: Increased Risk of Local Recurrence. Ann Surg. 2022 Feb 1;275(2):e420-e427. doi: 10.1097/SLA.0000000000003889. PMID 32224742
- [Derived] Deijen CL, Vasmel JE, de Lange-de Klerk ESM, Cuesta MA, Coene PLO, Lange JF, Meijerink WJHJ, Jakimowicz JJ, Jeekel J, Kazemier G, Janssen IMC, Pahlman L, Haglind E, Bonjer HJ; COLOR (COlon cancer Laparoscopic or Open Resection) study group. Ten-year outcomes of a randomised trial of laparoscopic versus open surgery for colon cancer. Surg Endosc. 2017 Jun;31(6):2607-2615. doi: 10.1007/s00464-016-5270-6. Epub 2016 Oct 12. PMID 27734203
- [Derived] Colon Cancer Laparoscopic or Open Resection Study Group; Buunen M, Veldkamp R, Hop WC, Kuhry E, Jeekel J, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy A, Bonjer HJ. Survival after laparoscopic surgery versus open surgery for colon cancer: long-term outcome of a randomised clinical trial. Lancet Oncol. 2009 Jan;10(1):44-52. doi: 10.1016/S1470-2045(08)70310-3. Epub 2008 Dec 13. PMID 19071061